CLINICAL TRIAL: NCT04992572
Title: Randomized Study Comparing Local/ MAC Anesthesia to General for 1-3 Level Lumbar Decompressions
Brief Title: Study Comparing Local/ MAC Anesthesia in Lumbar Decompression
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Todd Alamin, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61453
Record Dates: First submitted 2021-07-21; First posted 2021-08-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Propofol; Lidocaine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- General anesthesia (Active Comparator): Patients under this group will be undergoing lumbar decompression surgery with general anesthesia:
  General Anesthesia: Medically induced unconsciousness that suppresses reflexes and requires intubation (a tube inserted through the mouth and into the airway) to assist in breathing.
  Interventions: Drug: Propofol Injection
- Monitored Anesthetic Care (MAC)/Local (Active Comparator): Patients under this group wil be undergoing limbar decompression surgery with Monitored Anesthetic care, (MAC)/Local.
  Local + MAC: Local anesthetic (lidocaine) injected into the site of the incision/dissection with additional IV medication (Propofol) to achieve a state in which the patient is generally aware, but relaxed.
  Interventions: Drug: Lidocaine Hydrochloride, Injectable

INTERVENTIONS:
Drug: Propofol Injection — 25mg Propofol administered by injection
  Arms: General anesthesia
Drug: Lidocaine Hydrochloride, Injectable — Licocaine administered locally via injection.
  Arms: Monitored Anesthetic Care (MAC)/Local

SUMMARY:
Explore efficacy, complications, and other factors associated with anaesthetic choice- To evaluate the efficacy of local + MAC as an alternative anesthetic to general anesthesia and to analyze patients' outcomes and experiences.

DETAILED DESCRIPTION:
100 Patients ages 40-95 with lumbar stenosis to be decompressed are randomized to undergo the procedure with either general anesthesia or local anesthetic with MAC.

Participants will be randomized to either group 1 General anesthesia or group 2 Local + MAC anesthetic group.

Group 1: General Anesthesia: Medically induced unconsciousness that suppresses reflexes and requires intubation (a tube inserted through the mouth and into the airway) to assist in breathing.

Group 2: Local + MAC: Local anesthetic (lidocaine) injected into the site of the incision/dissection with additional IV medication (Propofol) to achieve a state in which the patient is generally aware, but relaxed

ELIGIBILITY:
Inclusion Criteria:

Patients with lumbar stenosis to be decompressed over 1-3 segments

* Ages 40-95
* Appropriate for general anesthesia

Exclusion Criteria:

* Planned significant nerve root retraction
* Previous fusion operation
* Unable to comply with follow up
* Patients with daily morphine equivalents or more 100mg
* Patients with a known hypersensitivity to propofol or any of DIPRIVAN Injectable Emulsion components.
* Patients with allergies to eggs, egg products, soybeans or soy products.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) score | Basline through year 2
  Scale is expressed as a percentage (0 to 100%). Higher score indicates more severe disability.
Change in patient reported pain | Basline through year 2
  Measured on visual analog scale (VAS). Score range 0-10, 0= no pain and 10 = worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Alamin, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Outpatient Surgery Center/Stanford Spine Clinic, Redwood City, California
  - Stanford Outpatient surgery center, Redwood City, California

IPD SHARING:
Plan to Share IPD: No